CLINICAL TRIAL: NCT01458002
Title: Online Tailored Interventions & Relational Agents for Exercise and Sun Protection
Acronym: Project RAISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rhode Island (Other)
Collaborators: Northeastern University (Other); Pro-Change Behavior Systems (Other)
Responsible Party: Principal Investigator, Wayne F. Velicer, Professor, University of Rhode Island
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: CA119195
Record Dates: First submitted 2011-09-20; First posted 2011-10-24 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Sedentary; Skin Cancer
MeSH Terms: conditions — Sedentary Behavior; Skin Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Assessment only
- Tailored Internet Communications (Other): TTM expert system only
  Interventions: Other: Tailored Internet Communication with Relational Agent; Other: Tailored Internet Communications
- Tailored Internet Communication with Relational Agent (Experimental): TTM expert system plus relational agent
  Interventions: Other: Tailored Internet Communication with Relational Agent

INTERVENTIONS:
Other: Tailored Internet Communication with Relational Agent — The Tailored Internet Intervention will include a "relational agent" component, which is an animated conversational agent that builds a working relationship with subjects over time and uses this alliance to boost intervention effectiveness and retention to the Tailored Internet Communications web site.
  Arms: Tailored Internet Communication with Relational Agent; Tailored Internet Communications
Other: Tailored Internet Communications — Best practices for TTM tailored communications with two types of feedback: normative - compared to peers and ipsative - self compared to previous assessment.
  Arms: Tailored Internet Communications

SUMMARY:
This study targets two major risk factors for cancer; is designed to treat the behaviors on a population basis, using proactive recruitment strategies; intervenes on multiple behaviors simultaneously, thereby producing greater impacts for cancer prevention; utilizes one of the most promising approaches to low cost population based interventions for health-related behavior change, namely the internet; and develops and tests a promising new approach to increasing the utilization and effectiveness of internet-based interventions, relational agents. The primary aims are: (1) To develop and assess the effectiveness of a tailored internet intervention on a national sample; (2) To develop and assess the effectiveness of the internet intervention enhanced by a relational agent; and (3) To determine if the intervention with the relational agent can outperform the regular tailored internet intervention.

DETAILED DESCRIPTION:
The overarching goal of this research project is to revise and enhance a multimedia computer-based multiple risk factor intervention for cancer prevention, using the internet to reach a general population. Two innovative, individualized, easily disseminated, low-cost, and interactive interventions, both for multiple behaviors (sun protection and exercise adoption), will be developed and evaluated in comparison to a control condition. The first intervention involves adapting our effective multimedia expert system interventions to the internet environment. The second intervention builds on the first with the additional inclusion of a Relational Agent, a recently developed computer-based approach to establishing a personal relationship typically missing on internet sites. Both systems will employ the same theoretical model of behavior change, the Transtheoretical Model, as the deep knowledge, and all systems will employ empirically based decision rules. The design is a 3 Group (Control, Internet, Internet plus Relational Agent) x 3 Occasions (0, 12, 24 • Months) with intervention occurring during the first 12 months. A representative national sample of 1639 individuals at risk for both behaviors will be recruited. The primary aims are: (1) To develop and assess the effectiveness of a tailored internet intervention on a national sample; (2) To develop and assess the effectiveness of the internet intervention enhanced by a relational agent; and (3) To determine if the intervention with the relational agent can outperform the regular tailored internet intervention. The secondary aims are: (1) To determine if the two interventions are differentially effective with each behavior and with different subgroups, and (2) To determine if the relational agent intervention is utilized more often for increasing exercise than for sun protection. This study targets two major risk factors for cancer; is designed to treat the behaviors on a population basis, using proactive recruitment strategies; intervenes on multiple behaviors simultaneously, thereby producing greater impacts for cancer prevention; utilizes one of the most promising approaches to low cost population based interventions for health-related behavior change, namely the internet; and develops and tests a promising new approach to increasing the utilization and effectiveness of internet-based interventions, relational agents.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* access to computer
* willing to download materials

Exclusion Criteria:

* heart attack in past 6 months
* kidney failure during dialysis
* currently receiving chemotherapy or radiation for cancer
* had a seizure in the past 6 months
* had a leg or pelvic fracture in the past 6 months
* legally blind
* regularly use a wheelchair
* (women only) currently pregnant or plan to be pregnant in the next 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1364 (Actual)
Dates: Start 2009-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Exercise | Percentage of baseline at-risk participants who reach the Regular Exercise criteria at 24 months.
  Regular Exercise is defined as any planned physical activity (e.g., brisk walking, aerobics, jogging, bicycling, swimming, rowing, basketball, etc.) performed to increase physical fitness. Such activity should be performed 5 times or more per week for 30 minutes per session, consistent with CDC guidelines.
Sun Exposure | Percentage of baseline at-risk participants who reach the Sun Protection criteria at 24 months
  Consistently protecting themselves from the sun every time they were out in the sun for 15+ minutes is defined as 1) using sunscreens with a sun protection factor (SPF) of 15 or more, wearing protective clothing (for example, a hat with a wide brim, shirts, and pants), and avoiding or limiting exposure to the sun during the mid-day hours (10 am - 4 pm).

SECONDARY OUTCOMES:
Exercise | Increase in number of minutes of physical activity per week (150 minutes of moderate intensity or 75 minutes of vigorous intensity) measured by the International Physical Activity Questionnaire (IPAT)
Sun Exposure | Increase in number of sun protection behaviors as measured by the Sun Protection Behavior Scale (SPBS), which consists of three scales: sunscreen use, sun avoidance and protective clothing, and hat use.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne F Velicer, PhD, Principal Investigator — Univeristy of Rhode Island
Locations (1):
- University of Rhode Island, Kingston, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Redding CA, Prochaska JO, Paiva A, Rossi JS, Velicer W, Blissmer BJ, Greene GW, Robbins ML, Sun X. Baseline stage, severity, and effort effects differentiate stable smokers from maintainers and relapsers. Subst Use Misuse. 2011;46(13):1664-74. doi: 10.3109/10826084.2011.565853. Epub 2011 Mar 30. PMID 21449711